CLINICAL TRIAL: NCT00109135
Title: A Double-Blind, Multicenter, Randomized, Titrated-Dose, Placebo-Controlled, Study of MK0364 (4 mg to 8 mg) in Chronic Cigarette Smokers as an Aid for Smoking Cessation
Brief Title: A Study to Investigate a Research Drug as an Aid for Smoking Cessation in Chronic Cigarette Smokers (0364-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0364-007; 2005_012; MK-0364-007
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — N-(3-(4-chlorophenyl)-2-(3-cyanophenyl)-1-methylpropyl)-2-methyl-2-((5-(trifluoromethyl)pyridin-2-yl)oxy)propanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: taranabant
  Other Names: MK0364

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of an investigational drug that may help individuals to stop smoking.

ELIGIBILITY:
Inclusion Criteria:

* Smoking greater than/equal to 10 cigarettes/day for at least 1 year
* Laboratory tests that meet the criteria of the study
* In overall good health as determined by the investigator

Exclusion Criteria:

* Psychiatric diagnoses
* Certain cancers
* Patients who use nicotine replacement therapy
* Patients on a diet regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Quitting smoking after 8 weeks of treatment by measuring lab values and expired breath CO levels | after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director

REFERENCES:
- [Derived] Morrison MF, Ceesay P, Gantz I, Kaufman KD, Lines CR. Randomized, controlled, double-blind trial of taranabant for smoking cessation. Psychopharmacology (Berl). 2010 Apr;209(3):245-53. doi: 10.1007/s00213-010-1790-2. Epub 2010 Feb 27. PMID 20191360